CLINICAL TRIAL: NCT00795392
Title: Preoperative Psychological Evaluation as Predictor of Post-surgical Outcomes
Brief Title: Preoperative Psychological Evaluation as Predictor of Outcomes
Acronym: PEPO
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Other Study IDs: NJMU200811010; NJFY0811008
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Elective Surgery
Keywords: Psychology; Postoperative outcome; Surgical Operation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients assessed with ASA physical status scale
  Interventions: Other: ASA scale
- 2: Patients assessed with full-scale psychological factors
  Interventions: Other: Full-scale psychological assessment

INTERVENTIONS:
Other: ASA scale — ASA scale evaluation before operation
  Groups: 1
Other: Full-scale psychological assessment — Full-scale psychological evaluation before operation
  Groups: 2

SUMMARY:
Perioperative psychological care is increasingly recognized as an essential part in the surgical environment. Previous studies have developed a strategy to evaluate the psychological influence after operations and found that postoperative psychological states significantly associated with the outcomes of patients. However, preoperative evaluation of patients the physicians do thus far is mainly the physical status assessment following the scale of American Society of Anesthesiologists (ASA). Whether a full-scale evaluation of preoperative psychological status to surgical patients could be a predictor to postoperative outcomes or not is not still completely understood. The investigators hypothesized that the preoperative psychological assessment would be an important predictor to outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgical operation
* Age from 18-65 years

Exclusion Criteria:

* Age <18 years or >65 years
* Not willing to participate in this study
* Patients from emergency department

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All types of patients undergoing surgical operations
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Time of recovery | Since the end of the operation (1 day) to six-month follow-up.

SECONDARY OUTCOMES:
Intraoperative consumption of drugs | From the time of start of operation (0 min) to the end of the surgical procedures, this time will undergo alteration in different individuals
Hospitalization days | Time length of staying at hospital from the day of inpatient to discharge home, this time will undergo alteration in different individuals
Life quality | Since the end of the operation (1 day) to six-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China